CLINICAL TRIAL: NCT06990711
Title: A Phase 1 Clinical Trial of Siltuximab for the Treatment of Antibody-Mediated Rejection After Lung Transplantation (Siltux-AMR)
Brief Title: A Phase 1 Clinical Trial of Siltuximab for the Treatment of Antibody-Mediated Rejection After Lung Transplantation
Acronym: Siltux-AMR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Derek E Byers, MD, PhD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SILTUX_AMR2025; 7R61HL169189-02 (NIH)
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Antibody Mediated Rejection of Lung Transplant
Keywords: lung transplant; antibody mediated rejection; transplant rejection; IL-6 blockade; donor specific antibodies
MeSH Terms: interventions — siltuximab

STUDY DESIGN:
Intervention Model Description: Randomized 1:1:1
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Siltuximab full-dose (11mg/kg) IV (Experimental): Siltuximab 11mg/kg IV on Days 1 and 22
  Interventions: Drug: Siltuximab
- Siltuximab half-dose (5.5mg/kg) IV (Experimental): Siltuximab 5.5 mg/kg IV on Days 1 and 22
  Interventions: Drug: Siltuximab
- Placebo IV (Placebo Comparator): Placebo IV on Days 1 and 22
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Siltuximab — Interleukin-6 blockade
  Arms: Siltuximab full-dose (11mg/kg) IV; Siltuximab half-dose (5.5mg/kg) IV
Drug: Placebo — Siltuximab placebo IV
  Arms: Placebo IV

SUMMARY:
Antibody-mediated rejection after lung transplantation commonly results in allograft failure and death in spite of current therapeutic regimens. We are testing the safety and tolerability of the addition of a novel immunosuppressive medication to routine treatment for antibody-mediated rejection. Future studies will be needed to assess efficacy if this study demonstrates safety

DETAILED DESCRIPTION:
Long-term outcomes after lung transplantation remain disappointing, and the median survival is 6.7 years. Chronic lung allograft dysfunction (CLAD) is the leading cause of death beyond the first year after lung transplantation. Antibody-mediated rejection (AMR), which is increasingly recognized after lung transplantation, is caused by donor-specific antibodies (DSA) to mismatched human leukocyte antigens (HLA) and frequently results in CLAD and death. Recent multicenter studies using intensive monitoring for AMR report an incidence over 25%. Treatment for AMR has generally focused on antibody depletion and prevention of additional antibody development. Various combinations have been used including high-dose corticosteroids, intravenous immune globulin (IVIG), Rituximab, Carfilzomib, anti-thymocyte globulin (ATG), and plasma exchange (PLEX). However, there have been no randomized controlled trials to guide management, and outcomes after AMR are dismal. One-year allograft survival after AMR is approximately 50%, and 2-year survival is only 20%. IL-6, initially identified as B-cell stimulating factor 2 (BSF-2), is a pleiotropic cytokine that drives deleterious inflammatory, alloimmune, and fibrogenic responses. In conjunction with other cytokines, IL-6 is responsible for normal antibody production and is critical for the induction of follicular helper T cells as well as the production of IL-21 which regulates immunoglobulin synthesis. IL-6 is also crucial for B-cell differentiation into plasmablasts and for enhancing plasmablast survival. These characteristics make IL-6 an especially attractive cytokine to target in the management of AMR. Human studies examining the role of IL-6 signaling blockade in the management of AMR after kidney transplantation have shown promising results, even in refractory cases. Preliminary experience with use of IL-6 signaling blockade in a very small number of lung transplant recipients with AMR has been encouraging. The principal hypothesis for this study is that IL-6 signaling blockade added to routine immunosuppressive treatment for AMR will improve clinical outcomes. However, evaluating the safety of this approach is necessary before examining efficacy in larger clinical trials because infections are the most common serious adverse events associated with IL-6 signaling blockade and a common cause of death at all timepoints after lung transplantation. This study is a Phase 1 clinical trial using Siltuximab, a monoclonal antibody to IL-6, in addition to routine immunosuppressive therapy for AMR to examine safety and define the optimal dose for the treatment of AMR. The primary endpoint is safety and tolerability, and secondary endpoints include pharmacodynamics and functional biological measures relevant to AMR (e.g., DSA, cell-free DNA). Data from this trial will inform the design of a future Phase 2 clinical trial that assesses efficacy. Carefully designed and implemented clinical trials are necessary to improve outcomes after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older,
2. Single or bilateral lung transplant recipient,
3. New diagnosis of clinical definite, probable, or possible antibody-mediated rejection according to the 2016 International Society for Heart and Lung Transplantation (ISHLT) definition with plans to be treated with Carfilzomib and/or anti-thymocyte globulin,
4. Admitted to the hospital for treatment of AMR,
5. Donor-specific antibodies (DSA) to human leukocyte antigens (HLA) with a Mean Fluorescence Intensity (MFI) > 1000,
6. Able to understand the purpose of the study and willing to participate and sign informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding,
2. Airway anastomotic dehiscence on bronchoscopy,
3. Thoracotomy incision dehiscence,
4. Underwent lung transplantation less than 6 months before enrollment,
5. Treated with rabbit anti-thymocyte globulin (ATG) for induction immunosuppression at the time of lung transplantation,
6. Underwent other invasive surgical procedure less than 6 weeks before enrollment,
7. History of lymphoma or hematologic malignancy,
8. Treatment with IL-6 signaling blockade with 6 months of enrollment,
9. Planned treatment with plasma exchange (PLEX) for AMR,
10. Cancer other than non-melanoma skin cancer with disease-free period < 3 years,
11. Positive respiratory virus PCR detected within 7 days of enrollment,
12. Active cytomegalovirus infection within 7 days of enrollment,
13. Positive respiratory culture for Mycobacterium tuberculosis, Mycobacterium abscessus, Mycobacterium chelonae, or Mycobacterium avium complex within 4 weeks of enrollment,
14. Absolute neutrophil count (ANC) < 1,000 cells/mm3 at enrollment,
15. Platelet count < 75,000 cells/mm3 at enrollment,
16. Hemoglobin ≥ 17 g/dL at enrollment,
17. ALT or AST > 2.5 times upper limit of normal at enrollment,
18. Total bilirubin > 2.5 times upper limit of normal at enrollment,
19. Uric acid ≥ 7 mg/dL at enrollment.
20. History of gastrointestinal tract perforation,
21. History of diverticulitis (diverticulosis is not an exclusion),
22. Plan for surgical procedure (other than bronchoscopy) within 120 days of enrollment.
23. Inability or unwillingness to give written informed consent or comply with the study protocol,
24. Any condition that in the opinion of the site investigator introduces undue risk by participating in this study or impacts the quality or interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of CTCAE ≥ grade 3 | From Randomization to Day 90.
  The primary objective is to assess the safety and tolerability of Siltuximab added to routine immunosuppressive treatment for AMR after lung transplantation. The dose of siltuximab (11mg/kg or 5.5 mg/kg) with the least side effect profile will be use for future trials of siltuximab in antibody mediated rejection in lung transplantation.

SECONDARY OUTCOMES:
incidence of CTCAE ≥ grade 3 | during a period of 180 days after randomization
serum high-sensitivity CRP | Up to 90 and 180 days after randomization
  Pharmacodynamic measure of Il-6 pathway blockade.
Blood Sultiximab levels | Up to 90 days after randomization
  pharmacokinetic measure
Clearance of donor specific antibodies | From randomization to day 180
Infections | Between randomization and day 180
  Confirmed bacterial, CMV (defined as a positive blood viral load ≥ 200 IU/mL), mold, mycobacterial, community-acquired respiratory viral infection (each assessed independently), or other opportunistic infection
Change in Forced Vital Capacity (FVC) | between randomization and day 180
Change in Forced Expiratory Volume in One Second (FEV1) | between randomization and day 180
Development of Chronic Lung Allograft Dysfunction | between randomization and day 180
  Development of probable CLAD according to the 2019 ISHLT criteria
Allograft survival | between randomization and day 180
  Allograft survival defined as death or undergoing re-transplantation
Hyperuricemia | between randomization and day 180
  Blood uric acid > 7 mg/dL
Hyperlipidemia | between randomization and day 180
  Hyperlipidemia requiring the initiation or dose increase of medical therapy

OTHER OUTCOMES:
Donor-derived cell-free DNA < 1% | up to day 180
Change in circulating donor-derived cell-free DNA | up to day 180
Change in high-sensitivity CRP | between randomization and day 180
Serum IL-6 | at enrollment
  Serum IL-6 levels at enrollment only before administration of the first dose of Siltuximab
Exhaled breath condensate IL-6 | at enrollment
IL-6 bioavailability | Multiple timepoints between randomization and day 180.
  Serial measurements of IL-6 bioavailability by reporter gene assay (RGA).

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey Hachem, MD, Principal Investigator — University of Utah; Derek Byers, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School, of Medicine, Barnes-Jewish Hospital, St Louis, Missouri
  - University of Utah, Saint Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
final determination pending